CLINICAL TRIAL: NCT01470976
Title: Randomized Controlled Trial of Goal-directed Resuscitation in High-risk Patients Undergoing Cardiac Surgery
Brief Title: Goal-directed Resuscitation in High-risk Patients Undergoing Cardiac Surgery
Acronym: GRICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar, Supervisor of the Surgical Intensive Care Unit of the Heart Institute, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0565/11
Record Dates: First submitted 2011-10-17; First posted 2011-11-11 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Perioperative Hemodynamic Optimization; Cardiac Surgery
Keywords: Goal-directed therapy; Hemodynamic optimization; Cardiac surgery
MeSH Terms: interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal-directed Therapy (GDT) Protocol (Active Comparator)
  Interventions: Other: Goal-directed Resuscitation Therapy (GDT)
- Standard Protocol (Active Comparator)
  Interventions: Other: Standard protocol

INTERVENTIONS:
Other: Goal-directed Resuscitation Therapy (GDT) — * A target value of a cardiac index (CI) greater than 3.0 L/min/m2 will be sought.
  * The first step will be fluid resuscitation with 250ml aliquots of Lactated Ringer's solution whenever the CI is lower than 3,0 L/min/m2 and systolic volume index (SVI) is lower than 35ml/m2. The fluid challenge will be stopped if the CVP rises by more than 4 mmHg during the infusion period.
  * When the CI is lower than or equal to 3,0L/min/m2 and SVI higher than or equal to 35 ml/m2, dobutamine will be initiated with increasing doses up to 20mcg/kg/min.
  * The final step will be red blood transfusion to reach a hematocrit higher than 28%.
  Other Names: LiDCO Rapid will be used to calculate CI and SVI.
  Arms: Goal-directed Therapy (GDT) Protocol
Other: Standard protocol — The control group will be managed by the anesthetic team in the operative room and by the surgical ICU staff in the postoperative period according to institutional protocol of hemodynamic monitoring.
  Arms: Standard Protocol

SUMMARY:
The primary aim of the study is to investigate whether a goal-directed resuscitation therapy in high-risk patients through cardiac index optimization using the LiDCO Rapid device reduces complications after cardiac surgery. The hypothesis is that there are better outcomes when achieving a cardiac index higher than 3L/min/m2 in those patients with an arterial lactate higher than 1.5 mmol/L.

ELIGIBILITY:
Inclusion Criteria:

* All elective primary and redo adult cardiac surgical patients for coronary artery bypass grafting, valve procedure or combined procedures
* Adults patients
* Written informed consent
* One of the following criteria:

  * EuroSCORE (European System for Cardiac Operative Risk Evaluation) higher than or equal to 6
  * Ejection fraction lower than 50%
  * Recent myocardial infarction
  * Unstable angina

Exclusion Criteria:

* Age less than 18 years
* Infectious endocarditis
* Transplant procedures
* Emergency procedures
* Pulmonary hypertension
* Preoperative cardiogenic shock or use of dobutamine
* Congenital procedures
* Need for intra-aortic balloon pump (IABP)
* Noradrenaline dose higher than 1mcg/kg/min
* Pregnancy
* Patients who refused participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Composite of death or major postoperative complications | within 30 days after cardiac surgery
  Death or one of the following complications: stroke, renal failure, respiratory complications, cardiovascular complications, deep wound infection and reoperation for any reason.

SECONDARY OUTCOMES:
Duration of ICU stay and hospital stay. | within 30 days after cardiac surgery
  To compare the number of days of ICU stay and hospital stay between groups.
Tissue hypoperfusion markers | within 30 days after cardiac surgery
  To compare levels of DO2, lactate, ScvO2, base excess and venous to arterial carbon dioxide difference between groups.
Cardiovascular measures | within 30 days after cardiac surgery
  To compare levels of BNP, myocardial enzymes, echocardiographic measures and free-days of vasopressors and inotropes between groups.
Mechanical ventilation | within 30 days after cardiac surgery
  To compare the number of mechanical ventilation free-days between groups.
Fluid balance | during ICU stay
  To compare fluid balance during ICU stay between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ludhmila A Hajjar, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto do Coracao - InCor / HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Hajjar LA, Fukushima JT, Osawa E, Almeida JP, Galas FR. Dobutamine administration in patients after cardiac surgery: beneficial or harmful? Crit Care. 2011;15(5):444. doi: 10.1186/cc10439. Epub 2011 Sep 27. No abstract available. PMID 21958463
- [Background] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381